CLINICAL TRIAL: NCT03853694
Title: A Multicenter, Randomized, Active-Controlled Study to Evaluate the Efficacy and Safety of EXPAREL When Administered Via Infiltration Into the Transversus Abdominis Plane Versus Standard of Care in Subjects Undergoing Elective Cesarean Section (CHOICE)
Brief Title: Efficacy and Safety of EXPAREL Versus Standard of Care (SoC) in Subjects Undergoing Elective Cesarean Section
Acronym: CHOICE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 402-C-414
Record Dates: First submitted 2018-09-19; First posted 2019-02-26 (Actual); Results first posted 2022-07-18 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Elective Cesarean Section; Pain Management
Keywords: bupivacaine; EXPAREL; analgesic; TAP Block; C-Section; Cesarean Section; elective c-section; TAP
MeSH Terms: conditions — Agnosia | interventions — Morphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Standard of Care Group) (Active Comparator): 150 mcg Duramorph® + postoperative multi-modal pain regimen. No EXPAREL TAP infiltration
  Interventions: Drug: 150 mcg Duramorph + multi-modal pain regimen
- Group 2 (Duramorph + EXPAREL TAP) (Experimental): 50 mcg Duramorph + EXPAREL TAP infiltration + postoperative multi-modal pain regimen.
  Interventions: Drug: 50 mcg Duramorph+ EXPAREL + multi-modal pain regimen
- Group 3 (EXPAREL TAP) (Experimental): EXPAREL TAP infiltration + postoperative multi-modal pain regimen. No Duramorph.
  Interventions: Drug: Exparel TAP + multi-modal pain regimen

INTERVENTIONS:
Drug: 50 mcg Duramorph+ EXPAREL + multi-modal pain regimen — Intrathecal injection of 50 mcg Duramorph + EXPAREL administered via TAP infiltration + multi-modal pain regimen.
  Arms: Group 2 (Duramorph + EXPAREL TAP)
Drug: 150 mcg Duramorph + multi-modal pain regimen — Intrathecal injection of 150 mcg Duramorph + multi-modal pain regimen.
  Arms: Group 1 (Standard of Care Group)
Drug: Exparel TAP + multi-modal pain regimen — EXPAREL administered via TAP infiltration + multi-modal pain regimen.
  Arms: Group 3 (EXPAREL TAP)

SUMMARY:
The purpose of this study is to compare total opioid consumption by subjects in different treatment groups.

Another purpose of this study is to assess how well EXPAREL works, collect any safety data and assess your satisfaction using EXPAREL.

DETAILED DESCRIPTION:
This is a Phase-4, multicenter, randomized, active-controlled study in approximately 182 adult women undergoing elective C-section. All subjects will remain in the hospital for up to 72 hours post surgery.

Subjects will be screened within 30 days prior to surgery. During the screening visit, subjects will be assessed for any past or present medical conditions that in the opinion of the investigator would preclude them from study participation.

After the Informed Consent Form (ICF) is signed, a medical history, surgical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, alcohol breath test and urine drug screen, and clinical laboratory tests (hematology and chemistry) will be performed.

On Day 1, prior to the C-section, eligible subjects will be randomized in a 1:1:1 ratio into one of the three treatment groups listed below:

* Group 1: 150 mcg Duramorph® (SOC arm)+ postoperative multi-modal pain regimen as defined in this protocol. No EXPAREL TAP infiltration following skin-incision closure.
* Group 2: 50 mcg Duramorph + EXPAREL TAP infiltration following skin-incision closure + postoperative multi-modal pain regimen as defined in this protocol.
* Group 3: EXPAREL TAP infiltration following skin-incision closure + postoperative multi-modal pain regimen as defined in this protocol. No Duramorph.

Rescue Medication will be provided, as needed, for all subjects.

Subjects will remain in the hospital for up to 72 hours after surgery.

Total opioid burden and Pain intensity scores using a 10 cm Visual Analog Scale (VAS) will be collected.

Daily pain intensity score (VAS) and all pain medications will be collected through Day 14.

A phone call will be made to each subject on Day 14 and Day 30.

ELIGIBILITY:
Inclusion Criteria:

1. Females 18 years of age and older at screening.
2. Term pregnancies of 37 to 42 weeks gestation, scheduled to undergo elective C-section.
3. American Society of Anesthesiology (ASA) physical status 1, 2, or 3.
4. Able to provide informed consent, adhere to the study visit schedule, and complete all study assessments.

Exclusion Criteria:

1. Subjects who, in the opinion of the study site principal investigator, have a high-risk pregnancy.
2. Subjects with a pregnancy-induced medical condition or complication.
3. Subjects with 3 or more prior C-sections.
4. Pre-pregnancy body mass index >50 kg/m2.
5. Allergy, hypersensitivity, intolerance, or contraindication to any of the study medications.
6. Planned concurrent surgical procedure with the exception of salpingo-oophorectomy or tubal ligation.
7. Severely impaired renal or hepatic function.
8. Subjects at an increased risk for bleeding or a coagulation disorder.
9. Concurrent painful physical condition that may require analgesic treatment in the postsurgical period for pain that is not strictly related to the surgery.
10. Clinically significant medical disease in either the mother or baby that, in the opinion of the investigator, would make participation in a clinical study inappropriate.
11. History of, suspected, or known addiction to or abuse of illicit drug(s), prescription medicine(s), or alcohol within the past 2 years.
12. Administration of an investigational drug within 30 days or 5 elimination half-lives of such investigational drug.
13. Previous participation in an EXPAREL study.
14. Any clinically significant event or condition uncovered during the surgery that might render the subject medically unstable or complicate the subject's postsurgical course.
15. Receives the epidural component of combined spinal epidural (CSE) anesthesia during the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2020-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nayana Nagaraj, MD, PhD, MPH, Study Director — Pacira Pharmaceuticals, Inc
Locations (18):
- United States (18):
  - Stanford University School of Medicine, Stanford, California
  - University of Florida- Gainesville, Gainesville, Florida
  - University of Florida college of Medicine - Jacksonville, Jacksonville, Florida
  - Clinical Research Prime, Idaho Falls, Idaho
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - St. Peter's University Medical Center, New Brunswick, New Jersey
  - Columbia University Medical Center/NY Presbyterian Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson Medical Center, Philadelphia, Pennsylvania
  - Magee-Women's Hospital of UPMC, Pittsburgh, Pennsylvania
  - The University of Texas Medical Branch, Galveston, Texas
  - Inova Health System, Falls Church, Virginia
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habib AS, Nedeljkovic SS, Horn JL, Smiley RM, Kett AG, Vallejo MC, Song J, Scranton R, Bao X. Randomized trial of transversus abdominis plane block with liposomal bupivacaine after cesarean delivery with or without intrathecal morphine. J Clin Anesth. 2021 Dec;75:110527. doi: 10.1016/j.jclinane.2021.110527. Epub 2021 Oct 6. PMID 34626927

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
Started | 56 | 56 | 55
Completed | 53 | 47 | 51
Not Completed | 3 | 9 | 4
Not completed — Protocol Violation | 3 | 5 | 3
Not completed — Delivered early | 0 | 1 | 0
Not completed — not suitable to proceed | 0 | 1 | 0
Not completed — difficult surgery | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP) | Total
Number analyzed (Participants) | 53 | 48 | 52 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.2 (4.67) | 34.1 (4.93) | 32.7 (5.03) | 33.3 (4.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 48 | 52 | 153
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 7 | 18
  Not Hispanic or Latino | 46 | 43 | 45 | 134
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 5 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 3 | 7 | 15
  White | 41 | 36 | 34 | 111
  More than one race | 1 | 1 | 0 | 2
  Unknown or Not Reported | 3 | 3 | 3 | 9
Region of Enrollment [Number; unit: participants]
  United States | 53 | 48 | 52 | 153
American Society of Anesthesiologists (ASA) Physical Status Classification [Count of Participants; unit: Participants] — ASA I: normal, healthy patient ASA II: mild systemic disease ASA III Severe systemic disease that is not life threatening ASA IV: Severe systemic disease that is a constant threat to life
  Participants
    ASA I | 2 | 0 | 3 | 5
    ASA II | 47 | 45 | 39 | 131
    ASA III | 4 | 3 | 10 | 17
Body Mass Index (pre-pregnancy) [Mean (Standard Deviation); unit: kg/m^2] | 31.69 (5.091) | 31.08 (5.181) | 32.23 (6.179) | 31.68 (5.490)

OUTCOME MEASURES:

1. Primary Outcome: Total Postsurgical Opioid Consumption Through 72 Hours
Description: To Compare total opioid consumption through 72 hours following EXPAREL infiltration into the Transversus abdominus plane (TAP) with SOC in subjects undergoing an elective C-section
Time Frame: Through 72 hours post-surgery
Measure: Least Squares Mean (Standard Error); unit: OMED mg
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
Number analyzed (Participants) | 53 | 47 | 51
OMED mg | 69.3 (1.15) | 36.1 (1.16) | 22.1 (1.16)

2. Secondary Outcome: Percentage of Opioid-free Subjects
Description: Percentage of opioid-free subjects. LS Means probability from the logistic regression with treatment, site, age, and height as explanatory variables.
Time Frame: through 72 hours or hospital discharge, whichever came first
Population: LS Means probability from the logistic regression with treatment, site, age, and height as explanatory variables.
Measure: Number; unit: percentage of participants, opioid free
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
Number analyzed (Participants) | 53 | 47 | 51
percentage of participants, opioid free | 22.4 | 28.8 | 30

3. Secondary Outcome: Severity of Itching (Numeric Rating Scale Score)
Description: Severity of itching (Numeric Rating Scale score from 0(being none)-10(being the worst))
Time Frame: through 72 hours after surgery
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
Number analyzed (Participants) | 50 | 44 | 48
score on a scale | 1.48 (0.161) | 0.94 (0.176) | 0.61 (0.167)

4. Secondary Outcome: Opioid Related Symptom Distress Scale Score (ORSDS)
Description: The Opioid-Related Symptom Distress Scale (ORSDS) is a 4-point scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 10 symptoms. The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS is the average of 10 symptom-specific scores. Each question will receive a score from 0-4 the composite score for each subject is the average of all scores. A higher score indicates a worse outcome.
Time Frame: through 72 hours after surgery
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
Number analyzed (Participants) | 53 | 47 | 51
score on a scale | 0.33 (0.055) | 0.23 (0.053) | 0.35 (0.051)

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events (SAEs) were recorded from the time the ICF was signed through Day 14.
Arm/Group | Group 1 (Standard of Care Group) | Group 2 (Duramorph + EXPAREL TAP) | Group 3 (EXPAREL TAP)
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/48 | 0/52
Serious Adverse Events (participants affected / at risk) | 2/53 | 2/48 | 2/52
Other Adverse Events (participants affected / at risk) | 43/53 | 41/48 | 30/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Standard of Care Group) (N=53) | Group 2 (Duramorph + EXPAREL TAP) (N=48) | Group 3 (EXPAREL TAP) (N=52)
Postpartum hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Abdominal wall hematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (Standard of Care Group) (N=53) | Group 2 (Duramorph + EXPAREL TAP) (N=48) | Group 3 (EXPAREL TAP) (N=52)
Abdominal distention (Gastrointestinal disorders) | 6 | 6 | 2
Constipation (Gastrointestinal disorders) | 6 | 2 | 7
Flatulence (Gastrointestinal disorders) | 2 | 0 | 4
Nausea (Gastrointestinal disorders) | 16 | 9 | 2
Vomiting (Gastrointestinal disorders) | 4 (7) | 2 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 1 | 4 | 2
Dizziness (Nervous system disorders) | 2 | 4 | 1
Headache (Nervous system disorders) | 3 | 1 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 25 (74) | 28 | 16
Pruritus generalised (Skin and subcutaneous tissue disorders) | 9 (20) | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results conducted at Site shall not be published before 1st multicenter publication by Sponsor but can proceed if there is no such publication ≤18 months after study completion/termination at all sites and all data have been received. Before submitting manuscript/materials to an outside person/entity, site shall give Sponsor 60 days to review and comment. Site shall, upon request, further delay publication/presentation for ≤120 days to allow Sponsor to protect its interests in Inventions.

DOCUMENTS (2):
  • Study Protocol (2019-02-07): https://cdn.clinicaltrials.gov/large-docs/94/NCT03853694/Prot_002.pdf
  • Statistical Analysis Plan (2020-03-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT03853694/SAP_001.pdf